CLINICAL TRIAL: NCT06053645
Title: The Weight of Cardiovascular Disease: A Prospective Pilot Study of Obese Adults With Cardiovascular Disease Evaluated in a Novel Cardiometabolic Clinic
Brief Title: The Weight of Cardiovascular Disease
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kyla M. Lara-Breitinger, Principal Investigator, Mayo Clinic
Other Study IDs: 23-003696
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to evaluate the impact of a cardiometabolic clinic on percent body weight loss, body mass index (BMI), and visceral adiposity distribution in obese adults with cardiovascular disease (CVD) at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30 kg/m2
* At least one of the following CVD: atrial fibrillation (AF), coronary artery disease (CAD), HFpEF (heart failure with preserved ejection fraction), HFrEF (heart failure with reduced ejection fraction), ACHD (adult congenital heart disease), or valvular heart disease
* Patients evaluated in the Cardiometabolic clinic
* Willingness to complete questionnaires/surveys
* Ability to complete monthly self-assessments at home

Exclusion Criteria:

* BMI <30 kg/m2
* Pregnancy or lactating women
* Hemodynamically unstable CVD
* Active malignancy
* Autoimmune or systemic inflammatory diseases
* Severe renal or hepatic failure
* Being considered unsafe to participate as determined by the study physician
* Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic medications, or other medications as determined by the study NP or physician
* Patients with active psychosis, mania, or substance use disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the cardiometabolic clinic at Mayo Clinic Hospital in Rochester, MN will be recruited for participation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percent body weight loss | 12 months
  Total percent body weight loss will be reported at 12 months based on the following formula: (Starting baseline weight minus current weight) / (starting baseline weight) x 100 equals % of body weight loss.
Change in Body Mass Index (BMI) | Baseline, 12 months
  Body Mass Index (BMI) will be calculated using the standard formula from participants' height and weight. BMI = (Weight in Pounds / (Height in inches x Height in inches)) x 703
Change in visceral adiposity distribution | Baseline, 12 months
  Change in visceral adiposity distribution measured using dual energy X-ray absorptiometry (DEXA).

SECONDARY OUTCOMES:
Change in Blood Pressure | Baseline, 12 months
  Measured in millimeters of mercury (mmHg)
Change in point of care glucose | Baseline, 12 months
  Change in estimated glucose value (mg/dl) obtained from point of care fingerstick testing.
Change in quality of diet | Baseline, 12 months
  Change in quality of diet will be assessed by the Mini-EAT (Eating Assessment Tool). The Mini-EAT is a 9 item questionnaire that asks subjects how often they eat different types of foods (e.g. fruits, vegetables, legumes, etc.). Subjects respond on a scale of "I do not eat it at all" to "6 or more servings per day." Higher scores on the Mini-EAT represent a better quality of diet.
Change in psychosocial distress as measured by Screening Tool for Psychological Distress (STOP-D) | Baseline, 12 months
  Psychosocial distress will be measured by the STOP-D survey. The STOP-D survey asks subjects to rate how often over the last 2 weeks they have felt depressed, anxious, stressed, angry, or lacking social support on a scale of 0-Not at all to 9-Severely. Each item is scored separately without a summed score for overall distress. Higher individual scores on the STOP-D items represent worse psychosocial distress.
Change in psychosocial distress as measured by Impact of Event Scale-Revised (IES-R) | Baseline, 12 months
  Psychosocial distress will be measured by the IES-R. The IES-R is a questionnaire which asks subjects to rate how distressed or bothered during the past seven days they have been by difficulties that people sometimes have after stressful life events. Responses can range from 0-Not at all to 4-Extremely. Items on the questionnaire are grouped into 3 subscales: Intrusion, Avoidance, and Hyperarousal with scores on each subscale being the mean item response of all items in that group, thus scores for each subscale also range from 0 to 4. Higher scores are indicative of more psychosocial distress following the specific life event of focus.
Change in psychosocial distress as measured by Adverse Childhood Experience (ACE) Questionnaire | Baseline, 12 months
  Psychosocial distress will be measured by the ACE Questionnaire. The ACE Questionnaire asks subjects various questions regarding life experiences from the first 18 years of life that may be considered adverse experiences (e.g. parental abuse, neglect, parental divorce, etc.). Subjects answer each question with a yes or no selection. The more questions answered yes represents worse psychosocial distress.
Change in functional aerobic capacity (VO2 Max) | Baseline, 12 months
  VO2 Max is measured as milliliters of oxygen per kilogram of body weight per minute (ml/kg/min) during cardiopulmonary exercise test
Change in artificial intelligence electrocardiogram (AI-ECG) age | Baseline, 12 months
  AI-ECG age is the subject's predicted age based on artificial intelligence analysis of electrocardiograms (ECGs).
Change in E/e' | Baseline, 12 months
  E/e' will be measured using transthoracic echocardiography (TTE). It is defined as the ratio of peak early diastolic mitral inflow velocity (E) and peak early diastolic mitral annular velocity (e') and will be used to assess left ventricular diastolic function.
Change in Peak Tricuspid Regurgitation (TR) Velocity | Baseline, 12 months
  Peak TR Velocity (m/s) will be measured using transthoracic echocardiography (TTE) to assess left ventricular diastolic function.
Change in Right Atrial (RA) Pressure | Baseline, 12 months
  RA pressure (mm Hg) will be measured by transthoracic echocardiography (TTE) to assess left ventricular diastolic function.
Change in Left Atrial (LA) volume index | Baseline, 12 months
  LA volume index (ml/m^2) will be measured by transthoracic echocardiography (TTE) to assess left ventricular diastolic function.
Change in physical activity | Baseline, 12 months
  Average number of steps a subject takes daily as collected by an Apple watch worn by subjects for the duration of the study.
Change in heart rate with detection of arrhythmia | Baseline, 12 months
  Average number of arrhythmias identified by an Apple watch worn by subjects for the duration of the study.
Change in cardio fitness | Baseline, 12 months
  Fitness level reported as high/above average/below average/low as collected by an Apple watch worn by subjects for the duration of the study.
Change in six-minute walk test | Baseline, 12 months
  Measurement (meters) of distance a person can walk on flat ground in 6 minutes collected by an Apple watch worn by subjects for the duration of the study.
Change in psychosocial distress as measured by the Weight Bias Internalization-Modified (WBIS-M) scale | Baseline, 12 months
  The WBIS-M is a 11-item instrument for measuring the extent to which overweight individuals think of themselves in terms of prevalent negative stereotypes about overweight and overweight individuals. Respondents can express their level of agreement on a 7-point Likert scale ranging from 'strongly disagree' (1) to 'strongly agree' (7). Items 1 and 9 need to be scored reversely. Scores are averaged to create a composite score and higher scores represent greater psychosocial distress.

CONTACTS AND LOCATIONS:
Overall Officials: Kyla Lara-Breitinger, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No